CLINICAL TRIAL: NCT07044037
Title: Analysis of Cerebrospinal Fluid in Patients With Cerebral Toxoplasmosis at CHSD (2004-2024)
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 0076_NEUROLOGIE
Record Dates: First submitted 2025-06-12; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Toxoplasmosis, Cerebral; Toxoplasmosis; Meningitis; HIV Infections; Cerebrospinal Fluid; Central Nervous System Infections
MeSH Terms: conditions — Toxoplasmosis, Cerebral; Toxoplasmosis; Meningitis; HIV Infections; Central Nervous System Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This study looks at patients who were treated for cerebral toxoplasmosis at CHSD between 2004 and 2024. It focuses on analyzing their cerebrospinal fluid (CSF) to better understand the biological signs of the disease. The goal is to see if CSF results can show signs of meningitis, even though it's not commonly reported, and to describe any co-infections, symptoms, brain imaging findings, and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

- Adult patients (age 18 years) hospitalized at CHSD between January 1, 2004 and March 31, 2024 for cerebral toxoplasmosis

Exclusion Criteria:

- Under 18 years ols

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients (aged 18 years and older) who were hospitalized at the Centre Hospitalier de Saint-Denis (CHSD) between January 1, 2004, and March 31, 2024, with a principal or significant associated diagnosis of cerebral toxoplasmosis.
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | From hospital admission to completion of diagnostic lumbar puncture and initial treatment (typically within the first 7 days of hospitalization).

CONTACTS AND LOCATIONS:
Locations (1):
- France, Saint-Denis, France, France